CLINICAL TRIAL: NCT05669209
Title: Etiology and Contributing Factors of Anemia Among Women of Reproductive Age at Kebribeyah District in the Somali Regional State, Ethiopia
Brief Title: Causes of Anemia Among Women of Reproductive Age
Status: Completed | Type: Observational
Sponsor: Ethiopian Public Health Institute (Other Government)
Collaborators: Oklahoma State University (Other); Addis Ababa University (Other)
Responsible Party: Principal Investigator, Desalegn Kuche, Researcher for nutrition, Ethiopian Public Health Institute
Other Study IDs: EPHI_IRB_410_2021_1
Record Dates: First submitted 2022-12-04; First posted 2022-12-30 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Anemia
Keywords: Etiology; Anemia; Hemoglobin; Women of reproductive age
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We will collect blood, urine, and stool samples from all study participants. We will analyze for genetic causes of anemia (hemoglobinopathies) from the blood samples collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the causes of anemia in women of reproductive age. The main questions it aims to answer are:

* What are the causes of anemia among women of reproductive age?
* What is the contribution of iron deficiency to overall anemia?
* What is the prevalence of hemoglobinopathies among women of reproductive age with anemia?

Participants will be asked to respond to the interview questions, and provide blood, urine, and stool samples.

DETAILED DESCRIPTION:
One-third of the global population is affected by anemia making it one of the major public health problems at the global level. Women of reproductive age are at risk for anemia. The prevalence of anemia reported in 2016 Ethiopian Demographic and Health Survey (EDHS) is a moderate public health problem at the national level, but it is a severe public health problem in the Somali regional state among women of reproductive age (WRA). The purpose of this study is to assess the etiology and determinant factors of anemia among women of reproductive age. A cross-sectional design will be employed for the current study. In the current study, the investigators will assess the causes and contributing factors for anemia and their relationship with anemia. Women of reproductive age 18-49 years old residing in the Kebribeyah district are the target population for this study. The sample size determined for the current study is 881. The Somali region was selected for the current study due to its highest prevalence of anemia (60.6%%) among women of reproductive age according to the EDHS 2016. Kerbribeyah district was selected from the Somali regional state. Simple random sampling was employed to select three kebeles (villages) from the available kebeles with no other nutrition interventions in the Kebribeyah district. Two enumerations areas (EAs) from each of the three kebeles will be selected by simple random sampling. The sample size determined will be allocated to three kebeles and two EAs within the Kebeles on probability proportional to size (PPS). The study participants will be selected by systematic random sampling from a list of participants in a sampling frame obtained by house-to-house listing. After obtaining written informed consent, the data will be collected from the selected participant in their homes. All study participants who take part in the current study will be interviewed. They will also provide blood, urine, and stool samples. The prevalence of anemia and iron status biomarkers are the primary outcomes for the current study. The participants will be tested for anemia by measuring hemoglobin concentration. In addition, a complete blood count (CBC) test will be done for all study participants. The current study will fill the evidence gap by identifying major causes and contributors to overall anemia among women of reproductive age in the Kebribeyah district. The researchers anticipate that determining the causes of anemia will be a crucial first step in tackling the high prevalence of anemia among women of reproductive age in the Somali regional state and beyond.

ELIGIBILITY:
Inclusion Criteria:

* age range 18-49 years
* Permanent resident in the selected kebele (have lived for at least six months) in the kebele (village).

Exclusion Criteria:

* Women below or above the age range 18-49 years
* All pregnant women
* Women who are severely ill and incapacitated.
* Non-permanent resident women in the kebele (village)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The participants are expected to have the same gender identity as their biological sex.
Study Population: Women of reproductive age who are living in Kebribeyah district are the target population for this study. All non-pregnant women in the age range of 18-49 years living in three selected kebeles within the Kebribeyah district will be the study population. Our sample will be selected by systematic random sampling from a list of eligible women in the sampling frame. When there are two eligible women in the same household, one woman will be selected randomly.
Sampling Method: Probability Sample
Enrollment: 881 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Anemia prevalence | Single blood sample collected for the cross-sectional baseline study throughout a month on average.
  Anemia is diagnosed when the hemoglobin concentration test result is less than 12g/dl.
Iron deficiency anemia | Single blood sample collected for the cross-sectional baseline study throughout a month on average
  Iron deficiency anemia is diagnosed when serum ferritin concentration is less than 15μg/L and hemoglobin concentration is less than 12g/dl.

SECONDARY OUTCOMES:
Socioeconomic Status (SES) | From the cross-sectional baseline study conducted throughout a month on average
  Socioeconomic status will be assessed by using principal component analysis (PCA) from socio-demographic information collected.

CONTACTS AND LOCATIONS:
Overall Officials: Masresha Tessema, PhD, Study Director — Ethiopian Public Health Institute (EPHI)
Locations (1):
- Ethiopian Public Health Institute, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) can be shared upon request and signing agreement between Ethiopian Public Health Institute and the interested party.

REFERENCES:
- [Background] Cintron-Garcia J, Guddati AK. Effect of immigration on mortality trends in sickle cell patients. Am J Blood Res. 2020 Oct 15;10(5):172-178. eCollection 2020. PMID 33224561
- [Background] Daru J, Colman K, Stanworth SJ, De La Salle B, Wood EM, Pasricha SR. Serum ferritin as an indicator of iron status: what do we need to know? Am J Clin Nutr. 2017 Dec;106(Suppl 6):1634S-1639S. doi: 10.3945/ajcn.117.155960. Epub 2017 Oct 25. PMID 29070560
- [Background] Gebreegziabher T, Stoecker BJ. Iron deficiency was not the major cause of anemia in rural women of reproductive age in Sidama zone, southern Ethiopia: A cross-sectional study. PLoS One. 2017 Sep 12;12(9):e0184742. doi: 10.1371/journal.pone.0184742. eCollection 2017. PMID 28898272
- [Background] Kassebaum NJ, Jasrasaria R, Naghavi M, Wulf SK, Johns N, Lozano R, Regan M, Weatherall D, Chou DP, Eisele TP, Flaxman SR, Pullan RL, Brooker SJ, Murray CJ. A systematic analysis of global anemia burden from 1990 to 2010. Blood. 2014 Jan 30;123(5):615-24. doi: 10.1182/blood-2013-06-508325. Epub 2013 Dec 2. PMID 24297872
- [Background] Kibret KT, Chojenta C, D'Arcy E, Loxton D. Spatial distribution and determinant factors of anaemia among women of reproductive age in Ethiopia: a multilevel and spatial analysis. BMJ Open. 2019 Apr 4;9(4):e027276. doi: 10.1136/bmjopen-2018-027276. PMID 30948614
- [Background] Khambalia AZ, Aimone AM, Zlotkin SH. Burden of anemia among indigenous populations. Nutr Rev. 2011 Dec;69(12):693-719. doi: 10.1111/j.1753-4887.2011.00437.x. PMID 22133195
- [Background] Kohne E. Hemoglobinopathies: clinical manifestations, diagnosis, and treatment. Dtsch Arztebl Int. 2011 Aug;108(31-32):532-40. doi: 10.3238/arztebl.2011.0532. Epub 2011 Aug 8. PMID 21886666
- [Background] Liyew AM, Teshale AB. Individual and community level factors associated with anemia among lactating mothers in Ethiopia using data from Ethiopian demographic and health survey, 2016; a multilevel analysis. BMC Public Health. 2020 May 24;20(1):775. doi: 10.1186/s12889-020-08934-9. PMID 32448212
- [Background] Lopez A, Cacoub P, Macdougall IC, Peyrin-Biroulet L. Iron deficiency anaemia. Lancet. 2016 Feb 27;387(10021):907-16. doi: 10.1016/S0140-6736(15)60865-0. Epub 2015 Aug 24. PMID 26314490
- [Background] Petry N, Olofin I, Hurrell RF, Boy E, Wirth JP, Moursi M, Donahue Angel M, Rohner F. The Proportion of Anemia Associated with Iron Deficiency in Low, Medium, and High Human Development Index Countries: A Systematic Analysis of National Surveys. Nutrients. 2016 Nov 2;8(11):693. doi: 10.3390/nu8110693. PMID 27827838
- [Background] Teshale AB, Tesema GA, Worku MG, Yeshaw Y, Tessema ZT. Anemia and its associated factors among women of reproductive age in eastern Africa: A multilevel mixed-effects generalized linear model. PLoS One. 2020 Sep 11;15(9):e0238957. doi: 10.1371/journal.pone.0238957. eCollection 2020. PMID 32915880